CLINICAL TRIAL: NCT01336439
Title: Effects of Botulinum Toxin Type A(Meditoxin®) on Sleep Bruxism by Different Injection Sites Evaluated by Polysomnography
Brief Title: Effects of Botulinum Toxin Type A(Meditoxin®) on Sleep Bruxism
Acronym: BBP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Kim Seong Taek, Yonsei University dental hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2-2010-0017
Record Dates: First submitted 2011-04-04; First posted 2011-04-15 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Sleep Bruxism
Keywords: Bruxism; Polysomnography; Botulinum toxin type A; Masseter muscle; Temporal muscle
MeSH Terms: conditions — Sleep Bruxism; Bruxism | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- M group (Active Comparator): A total of 25U of botulinum toxin type A was injected into each side masseter muscle in this arm.
  Interventions: Drug: Botulinum toxin type A (Meditoxin®)
- MT group (Active Comparator): A total of 25U of botulinum toxin type A was injected into each side masseter and temporal muscle in this arm.
  Interventions: Drug: Botulinum toxin type A (Meditoxin®)

INTERVENTIONS:
Drug: Botulinum toxin type A (Meditoxin®) — In this study, the botulinum toxin type A (Meditoxin®)was supplied as a freeze-dried powder of 200U, and was reconstituted with 4ml of sterile saline to a concentration of 5U/0.1ml.
  After pre-injection polysomnography, botulinum toxin type A was injected into each side bilaterally using a 1ml-syringe with a 29-gauge, and a 1/2-inch needle. The "M group" had an injection in masseter muscle. The "MT group" had an injection in masseter and temporal muscle. A total of 25U of botulinum toxin type A was injected into each site.
  After 4 weeks, the subjects had a post-injection polysomnography.
  Other Names: Meditoxin®(PacificPharm corporation, Korea)

SUMMARY:
The purpose of this study is to evaluate the effect of Botulinum toxin type A(Meditoxin®) on bruxism using polysomnography and determine which site is most appropriate for injection to obtain maximal effects.

DETAILED DESCRIPTION:
Bruxism is an oral habit consisting of involuntary non-functional gnashing, clenching, grinding of teeth and is a very common condition in the general population. Various treatment modalities such as occlusal splints, pharmacologic agent and cognitive-behavioral therapy have been investigated for the management of bruxism, but none is reported to be fully effective. Recently locally injected botulinum toxin has been used in various movement disorders, but its usefulness and objective effects on nocturnal bruxism have not been evaluated using objective measures such as polysomnography. Moreover, there is no systematic study about which site is most appropriate for injection to obtain maximal effects.

The aim of this study is to evaluate the effect of botulinum toxin type A into masseter muscle or both masseter muscle and temporal muscle on nocturnal bruxism using polysomnography and the changes in the bruxism events on polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of sleep bruxism confirmed by wear facets on occlusal splint
* must be able to follow clinical trial procedure
* who are suitable for this clinical trial
* who participated in this clinical trial out of his own free will

Exclusion Criteria:

* who take medications such as benzodiazepine or muscle relaxants
* who have secondary bruxism due to brain injury
* who are pregnant or have the possibility of pregnancy
* who had an botulinum toxin injection during the past three months
* who had an allergic reaction history to botulinum toxin
* who have an infection or skin trouble on injection site
* who have an other treatment plan for bruxism
* who are enrolled in other clinical trials
* who are not suitable for this clinical trials
* who have mandibular dyskinesia or mandibular dystonia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The change of bruxism events | At 4 weeks after Botulinum toxin type A injection
  Before and after injection, we compared the change of bruxism event in polysomnography by sleep laboratory criteria.
  <Sleep laboratory criteria>
  - Mean SB EMG potential : >10% or 20% of the maximal clench while awake (masseter muscles)
  In M group, Botulinum toxin was injected into masseter muscle. In TM group, Botulinum toxin was injected into masseter muscle and temporal muscle.

SECONDARY OUTCOMES:
The change of masticatory force(%) | At 4 weeks after Botulinum toxin type A injection
  We evaluated the change of subjective masticatory force before and after the injection. We asked the subject that "when the masticatory force before injection is represented 100%, what the masticatory force after injection?"
The change of Pain | At 4 weeks after Botulinum toxin type A injection
  We asked the subject about change of pain if the subject has pain on masseter muscle due to myogeneous problem. Pain score was chosen from a scale of zero to 10, where zero represented 'no pain' and 10 represented 'the worst pain they had ever experienced' (Numerical rating scale, NRS)
Sleep-related movement disorders | At 4 weeks after Botulinum toxin type A injection
  The percentage of subjects who have sleep-related movement disorders(ex, Restless Legs Syndrome, Periodic Limb Movement Disorder, Sleep Related Leg Cramps, Sleep Related Rhythmic Movement Disorder Sleep Related Movement Disorder, Unspecified)except sleep related bruxism
Sleep-related breathing disorders | At 4 weeks after Botulinum toxin type A injection
  The percentage of subjects who have sleep-related breathing disorders(ex, Obstructive Sleep apnoea, Sleep Related Hypoventilation/Hypoxaemic syndromes, sleep Related Non-obstructive Alveolar Hypoventilation(idiopathic), Sleep apnoea/Sleep Related Breathing Disorder, Unspecified and etc.)

CONTACTS AND LOCATIONS:
Overall Officials: SeongTaek Kim, PhD, Study Chair — Yonsei University dental hospital
Locations (1):
- Yonsei University dental hospital, Seoul, Sedaemun-gu, South Korea